CLINICAL TRIAL: NCT05745792
Title: Clinico-immunological Characterization and Immune Tolerance Breakdown in HU-autoimmunity
Acronym: CarTo-Hu
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 751
Record Dates: First submitted 2023-02-12; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Immune Tolerance
Keywords: PARANEOPLASTIC NEUROLOGICAL DISORDERS; LUNG CANCER; HU AUTOIMMUNITY; IMMUNE TOLERANCE BREAKDOWN
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, PBMCs, DNA, CSF and tumor collected at the time of diagnosis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Hu Abs: Patients harboring Hu Abs and a neurological syndrome
  Interventions: Other: Description of clinical, immunological and tumor features of patients harboring Hu Abs

INTERVENTIONS:
Other: Description of clinical, immunological and tumor features of patients harboring Hu Abs — This observationnal study involves clinical data and bio. samples (DNA and tumors block). Demographic and clinical data already in French Reference Center on PNS database will be reviewed. Additional data will be obtained from the referral physicians. The results of diagnostic tests performed to detect Hu-Abs in the patients are already in this database and will be retrospectively analyzed. In addition, the 4 available techniques (immunofluorescence, commercial immunodot, Western blot, and CBA) will be performed from Jan. 2022 to Dec. 2022.Tumor samples from 2 cohorts will be analyzed: (i) tumors of patients with Hu-Abs and PNS, and (ii) tumors of patients without PNS (mostly SCLC). After selecting patients, the study will involve 3 steps: (i) pathological confirmation; (ii) DNA sequencing and CNV analysis (panel of genes involved in anti-Hu autoimmunity; mainly ELAVL1 to 4, encoding for HuA to HuD, the 4 main proteins of the Hu family); and (iii) whole-genome RNA sequencing.

SUMMARY:
Phenotypic characterization of patients with Hu-Abs, including the different neurological presentation and the presence or not of an underlying cancer.

Analysis and clinical correlation of the diagnostic techniques for Hu-Abs detection (immunofluorescence, immunodot/Western blot, and CBA) in serum and/or CSF.

Genomic and transcriptomic features of tumors (histological and immune infiltrate characteristics, transcriptomic profile, mutational status).

ELIGIBILITY:
* Inclusion Criteria * :

  * Patient with neurological disorder
  * Patient with Hu antibody in sera or CSF
* Exclusion Criteria * :

  * Patient with no data
  * Patient without neurological disorder
  * Patient without Hu antibody in sera/CSF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients harboring Hu Abs in serum and/or CSF with or without cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRs) | At 1 year
  Application of modified rankin scale

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites autoimmunes, Lyon, France